CLINICAL TRIAL: NCT00613002
Title: A Phase III, Randomized, Double-Blind, Placebo Controlled, Multi-Center Study of the Safety and Efficacy of LibiGel® for the Treatment of Hypoactive Sexual Desire Disorder in Surgically Menopausal Women
Brief Title: Safety and Efficacy of LibiGel® for the Treatment of Hypoactive Sexual Desire Disorder in Surgically Menopausal Women
Acronym: BLOOM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioSante Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TESTW006
Record Dates: First submitted 2008-01-30; First posted 2008-02-12 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: hypoactive sexual desire disorder; testosterone; menopause
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Testosterone Propionate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- testosterone gel (Experimental): 1% testosterone transdermal gel
  Interventions: Drug: testosterone gel
- placebo gel (Placebo Comparator): placebo transdermal gel
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: testosterone gel — once daily transdermal testosterone gel, 300 mcg
  Other Names: LibiGel
  Arms: testosterone gel
Drug: placebo gel — once daily transdermal placebo gel
  Arms: placebo gel

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multi-center study of the safety and efficacy of LibiGel® 300mcg in the treatment of HSDD in surgically menopausal women

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 30 to 65 years
* Must have undergone hysterectomy and bilateral salpingo-oophorectomy

Exclusion Criteria:

* A history of allergic reactions to androgens (oral or patch), topical alcohol, or any component of the formulation
* Any systemic skin diseases or local skin abnormalities in the area of application
* Diagnosed with another primary female sexual dysfunction (e.g., Sexual Aversion Disorder, Female Sexual Arousal Disorder).
* A medical condition that could affect or interfere with sexual function
* Using a systemic topical gel or cream estrogen therapy.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2006-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Co-primary endpoints are the change in the 4-week total number of satisfying sexual events from the Baseline period to Weeks 21-24, and the change from Baseline to Weeks 21-24 in the mean ISED desire score. | Baseline and 21-24 weeks.

SECONDARY OUTCOMES:
Change from baseline over time for multiple efficacy measurements | change over timepoints from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Snabes, MD, PhD, Study Director — BioSante Pharmaceuticals, Inc.
Locations (63):
- United States (60):
  - BioSante Site #215, Birmingham, Alabama
  - BioSante Site #095, Hoover, Alabama
  - BioSante Site #014, Huntsville, Alabama
  - BioSante Site #027, Glendale, Arizona
  - BioSante Site #040, Tucson, Arizona
  - BioSante Site #052, Hot Springs, Arkansas
  - BioSante Site #182, Buena Park, California
  - BioSante Site #008, San Diego, California
  - BioSante Site #007, Denver, Colorado
  - BioSante Site #216, Denver, Colorado
  - BioSante Site #036, Ridgefield, Connecticut
  - BioSante Site #013, Washington D.C., District of Columbia
  - BioSante Site #024, Miami, Florida
  - BioSante Site #219, Pinellas Park, Florida
  - BioSante Site #041, St. Petersburg, Florida
  - BioSante Site #009, West Palm Beach, Florida
  - BioSante Site #189, Addison, Illinois
  - BioSante Site #005, Shreveport, Louisiana
  - BioSante Site #004, Baltimore, Maryland
  - BioSante Site #044, Detroit, Michigan
  - BioSante Site #047, Grand Rapids, Michigan
  - BioSante Site #033, Saginaw, Michigan
  - BioSante Site #031, Saint Clair Shores, Michigan
  - BioSante Site #208, Edina, Minnesota
  - BioSante Site #198, Saint Paul, Minnesota
  - BioSante Site #051, Missoula, Montana
  - BioSante Site #006, Lincoln, Nebraska
  - BioSante Site #217, Las Vegas, Nevada
  - BioSante Site #015, Poughkeepsie, New York
  - BioSante Site #059, Cary, North Carolina
  - BioSante Site #079, Charlotte, North Carolina
  - BioSante Site #061, Winston-Salem, North Carolina
  - BioSante Site #056, Fargo, North Dakota
  - BioSante Site #210, Akron, Ohio
  - BioSante Site #212, Cincinnati, Ohio
  - BioSante Site #213, Columbus, Ohio
  - BioSante Site #050, Eugene, Oregon
  - BioSante Site #197, Wexford, Pennsylvania
  - BioSante Site #089, Columbia, South Carolina
  - BioSante Site #209, Greer, South Carolina
  - BioSante Site #097, Hilton Head Island, South Carolina
  - BioSante Site #038, Mt. Pleasant, South Carolina
  - BioSante Site #049, Watertown, South Dakota
  - BioSante Site #093, Bristol, Tennessee
  - BioSante Site #069, Chattanooga, Tennessee
  - BioSante Site #078, Memphis, Tennessee
  - BioSante Site #042, Nashville, Tennessee
  - BioSante Site #048, Austin, Texas
  - BioSante Site #073, Corpus Christi, Texas
  - BioSane Site #220, Dallas, Texas
  - BioSante Site #039, Houston, Texas
  - BioSante Site #211, San Antonio, Texas
  - BioSante Site #218, Murray, Utah
  - BioSante Site #096, Williston, Vermont
  - BioSante Site #003, Charlottesville, Virginia
  - BioSante Site #086, Norfolk, Virginia
  - BioSante Site #053, Richmond, Virginia
  - BioSante Site #090, Virginia Beach, Virginia
  - BioSante Site #083, Mountlake Terrace, Washington
  - BioSante Site #181, Tacoma, Washington
- Canada (3):
  - BioSante Site #188, Sarnia, Ontario
  - BioSante Site #054, Windsor, Ontario
  - BioSante Site #193, Shawinigan, Quebec

REFERENCES:
- See also: http://www.bloomstudy.com — http://www.bloomstudy.com